CLINICAL TRIAL: NCT01247701
Title: Umbilical Cord Blood Transplant for Children With Myeloid Hematological Malignancies (UCAML)
Brief Title: Umbilical Cord Blood Transplant for Children With Myeloid Hematological Malignancies
Acronym: UCAML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Caridad Martinez, Assistant Professor, Pediatric Hematology/Oncology, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26558-UCAML
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Myeloid Hematological Malignancies
Keywords: UCB; Umbilical Cord Blood; Transplant; Umbilical Cord Blood Transplant; Cord Blood Stem Cell Transplantation; Pediatric; Myeloid Hematological Malignancies; Busulfan; Cytoxan; Cyclophosphamide; Fludarabine
MeSH Terms: interventions — Busulfan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Blood Transplant (Experimental): Busulfan,Cyclophosphamide, Fludarabine, Cord Blood Stem Cell Infusion
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Cord Blood Stem Cell Infusion

INTERVENTIONS:
Drug: Busulfan — Busulfan dosing will be as follows: Patients < 12 kg: 1.1 mg/kg/dose IV every 6 hours for 16 doses total; patients > 12 kg: 0.8 mg/kg/dose IV every 6 hours for 16 doses. It will be given on Days -9, -8, -7 and -6.
  Other Names: Busulfex
Drug: Cyclophosphamide — Cyclophosphamide (50 mg/kg/dose) will be given IV on Days -5, - 4, -3, and -2 over 1 hour. The total dose to be given over 4 days is 200 mg/kg.
  Other Names: CTX, Cytoxan
Drug: Fludarabine — Fludarabine will be given IV daily over 1 hour for 3 days. Dosing will be as follows: for patients ≤ 10 kg: 1.3 mg/kg; for patients > 10 kg: 40 mg/m^2.
  Other Names: Fludera
Procedure: Cord Blood Stem Cell Infusion — The cord blood stem cells will be infused on Day 0.

SUMMARY:
In this study, the investigators will use busulfan and cyclophosphamide (BuCy) backbone with the addition of fludarabine as the preparative Stem Cell Transplant (SCT) regimen. As an attempt to improve engraftment rate and reduce infections, the investigators are going to incorporate fludarabine in the conditioning regimen. The use of a BuCy backbone has been widely used and comparable to total body irradiation and cyclophosphamide (Cy/TBI) regimen.

Encouraging data on adding fludarabine to the SCT regimen have been reported. A fludarabine-based, conditioning regimen, with adequate immunosuppressive activity could conceivably allow engraftment of stem cells from alternative donors in hematologic malignancies patients with acceptable engraftment rates and low transplant-related mortality. Regimen-related toxicity is believed to be a major contributing factor to GVHD. Therefore this approach may also lead to reduced GVHD, as some investigators have suggested.

In an attempt to decrease the rate of viral infection and reactivation, the investigators will avoid ATG (Thymoglobulin) / Campath (anti-CD52), and instead administer Mycophenolate Mofetil (MMF). The addition of fludarabine should compensate any increase risk of graft failure with the removal of the ATG/Campath. The investigators anticipate that the removal of ATG/Campath will facilitate immune reconstitution more efficiently after receiving a UCBT.

DETAILED DESCRIPTION:
The following will be given as the conditioning regimen for the transplant:

BUSULFAN: Busulfan (intravenous BUSULFEX) dosing will be as follows: patients <12 kg: 1.1 mg/kg/dose IV every 6 hours for 16 doses total; patients >12 kg: 0.8 mg/kg/dose IV every 6 hours for 16 doses. Administration and pharmacokinetic monitoring will be performed as per standard practice. Anticonvulsants will be given in accordance with standard Blood and Marrow Transplant Program recommendations.

CYCLOPHOSPHAMIDE: Cyclophosphamide (50 mg/kg/dose) will be given IV on Days -5, - 4, -3, and -2 over 1 hour. The total dose to be given over 4 days is 200 mg/kg. Mesna will be given in accordance with standard Blood and Marrow Transplant.

FLUDARABINE: Fludarabine will be given IV daily over 1 hour for 3 days. Dosing will be as follows: for patients ≤ 10 kg: 1.3 mg/kg; for patients > 10 kg: 40 mg/m2. Preparation, administration and monitoring will be according to standard practice procedure

POST-TRANSPLANT IMMUNOSUPPRESSION:

* CSA will begin on Day -3. For children < 40 kg, the initial dose will be 2.5 mg/kg IV over 2 hours every 12 hours. Dose adjustments will be made to maintain levels above 200 ng/mL. Levels will be done on Day 0 and then as clinical indicated. CSA will be tapered per institutional SOP. Once the patient can tolerate oral medications and has a normal gastrointestinal transit time, CSA will be converted to an oral form.
* MMF will begin on Day 0 at a dose of 15 mg/Kg IV or orally TID, and will be discontinued on Day +45 unless GVHD is present.

CNS Disease: Patients with CNS relapse or primary CNS disease that is symptomatic or associated to radiological changes will receive additional irradiation to the craniospinal axis.

SUPPORTIVE CARE:

* Supportive care will be provided as per standard practice of the Blood and Marrow Stem Cell Transplant program at the Texas Children's Hospital, including all prophylactic and therapeutic clinical care issues. These practices may be modified if necessary for any individual patient in order to provide optimum care for that particular patient.
* IVIG: Intravenous immunoglobulin (500 mg/kg per dose) will be given monthly until discontinuation of GVHD therapy and documentation of antibody production.
* CB-CTLs: Patients enrolled in this protocol may also be eligible for infusion of CB-derived multivirus-specific CTL to provide virus-specific immune reconstitution and treatment of viral infections after CBT.

EVALUATIONS DURING THE STUDY:

Screening Procedures; Pre-HCT:

* Physical examination
* Pregnancy test
* Complete blood count and chemistries
* Electrocardiogram
* Echocardiograph
* PT/PTT/Fibrinogen/Anti-Thrombin III/von Willebrand Factor
* Viral tests
* Bone marrow aspirate and biopsy/Lumbar puncture
* Renal Function (GFR)
* Lumbar puncture will be performed
* Pulmonary Function test

EVALUATIONS BETWEEN DAY 0 AND DAY 100:

* Physical examination
* Complete blood count and chemistries
* Lytes/BUN/Cr
* Peripheral blood for STRs or FISH analysis for molecular diagnostics
* Lymphocyte phenotype testing and lymphoproliferative responses
* Bone marrow aspirate and biopsy for assessment of leukemia status and UCB engraftment
* Lumbar puncture
* Immunoglobulins

EVALUATIONS AFTER DAY 100:

* Physical examination
* Complete blood count and chemistries
* Lytes/BUN/Cr
* Serum chemistries
* Peripheral blood with assessment of engraftment by STRs or FISH analysis and enzyme levels
* Echocardiograph with LVEF
* Bone marrow aspirate and biopsy assessment of leukemia status and UCB engraftment
* Lymphocyte phenotype testing (CD3, CD4, CD8, CD19 and CD56) and lymphoproliferative responses
* Immunoglobulins

FOLLOW-UP INTERVAL:

Patients will be seen in the hospital everyday until discharge. After discharge from the hospital, the patient will be following on the BMT clinics on a regular basis as recommended by the primary physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a myeloid hematologic malignancy (acute myelogenous leukemia, secondary myelogenous leukemia or myelodysplastic syndrome) unlikely to be cure by standard chemotherapy. This includes patients who have relapsed after standard chemotherapy treatments and patients in first remission with unfavorable prognostics features.
* Related or Unrelated Umbilical Cord Blood Unit with 0-1 antigen mismatch at HLA-A and B (at low resolution) and DRB1 (at high resolution), with a total nucleated cell dose of ≥ 4 x 10^7/kg.
* Lansky/Karnofsky scores at least 60.
* Written informed consent and/or signed assent line from patient, parent or guardian.
* Negative pregnancy test, if applicable.

Exclusion Criteria:

* Patients with uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections, patients must be receiving definitive systemic antifungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Severe renal disease (Creatinine > 3X normal for age).
* Severe hepatic disease (direct bilirubin > 3 mg/dL or SGOT > 500).
* Patient has DLCO < 50% predicted or FEV1 < 50% of predicted, if applicable.
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction < 20%).
* HIV positive.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caridad A Martinez, MD, Principal Investigator — Baylor College of Medicine; Robert A Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Umbilical Cord Blood Transplant
Started | 16
Completed | 6
Not Completed | 10
Not completed — Death | 2
Not completed — Relapsed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 1.5 [0.5 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 100 Days, 1 Year, and 3 Years After Umbilical Cord Blood Transplant in Pediatric Patients.
Description: To determine the overall survival rate at 1 year after umbilical cord blood transplant in pediatric patients with myeloid hematological malignancies.
Time Frame: 100 days, 1 year, and 3 years
Population: The analysis included all participants who enrolled in the study and underwent umbilical cord blood transplant (UCBT) except the one participant who died 4 days after transplant.
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 15
probability of overall survival
  100 days | 0.923 [0.566 to 0.989]
  1-Year | 0.923 [0.566 to 0.989]
  3-Year | 0.923 [0.566 to 0.989]

2. Secondary Outcome: Number of Participants With Severe Acute GVHD Grade III-IV
Description: Number of participants with acute GVHD graded by the method of Przepiorka et al, which evaluates skin involvement, lower and upper GI, and liver function (bilirubin), each being graded in stages from 0 to 4, where 0 means no acute GVHD, and 4 is the highest stage of acute GVHD.
Time Frame: Day 100
Population: The analysis included all participants who underwent Umbilical Cord Blood Transplant (UCBT) and were evaluable for acute GVHD. A participant was evaluable for acute GVHD if he/she engrafted and either completed 100 days observation after transplant or experienced acute GVHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 15
Participants | 2

3. Secondary Outcome: Number of Participants With Chronic GvHD
Description: Number of participants with chronic GVHD graded by the method of Przepiorka et al, which evaluates skin, joints, oral, ocular, hepatic, esophagus, GI, respiratory, platelet, and musculoskeletal involvement, in stages from 0 to 3.
Time Frame: 1 year
Population: The analysis included all enrolled participants who underwent umbilical cord blood transplant (UCBT) and were evaluable for chronic GVHD. A participant was evaluable for chronic GVHD if he/she engrafted and survived or remained in the study for more than 100 days after transplant. However, if the participant(s) relapsed within or around 100 days, they would not be evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 10
Participants | 1

4. Secondary Outcome: Number of Participants With Relapse Rate After Transplant
Description: To assess relapse rate at 1 and 3 years after transplant. Cumulative incidence of relapse was calculated from the date of umbilical cord blood transplant using the competing risk method as described in Gray(1988) with death prior to relapse as the competing risk. Participants still alive without a date of relapse were censored at the time of the last follow-up.
Time Frame: 1 and 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 15
percentage of participants
  1 year | 53.3 [24.8 to 75.3]
  3 year | 53.3 [24.8 to 75.3]

5. Secondary Outcome: Number of Participants With Donor Engraftment After Transplant.
Description: To evaluate donor engraftment at 100 days, 6, 9, 12, 24, and 36 months after transplant.
Time Frame: 100 days, 6, 9, 12, 24 and 36 months
Population: The analysis included all participants who underwent umbilical cord blood transplant (UCBT) except the one participant who died 4 days after transplant. If the participant(s) relapsed, they would not be evaluable for donor engraftment.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 12
Participants
  100 days | 11
  6 months: number analyzed (Participants) | 6
  6 months | 6
  9 months: number analyzed (Participants) | 6
  9 months | 6
  12 months: number analyzed (Participants) | 6
  12 months | 6
  24 months: number analyzed (Participants) | 6
  24 months | 6
  36 months: number analyzed (Participants) | 3
  36 months | 3

6. Secondary Outcome: Number of Participants With Platelet Engraftment
Description: Achievement of untransfused platelet count > 20 x 10^9/L on three consecutive days
Time Frame: Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 15
Participants | 13

7. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Achievement of absolute neutrophil count > 0.5 x 10^9/L on three consecutive days
Time Frame: Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 15
Participants | 15

ADVERSE EVENTS:
Time Frame: We have recorded all grade 3 and 4 toxicities, except hematological toxicities, fever, abnormal glucose, ALT, GGT, and K levels from the day conditioning started until day 30 post-transplant. SAEs were reported up to day 100. Our study primary outcome is Overall Survival (OS) up to 3 years after transplant. The use of AEs up to 100 days is the standard measurement after a stem cell transplant. OS will capture any major toxicity up to 3 years after transplant that will lead to mortality.
Description: The analysis included all participants who enrolled in the study and underwent umbilical cord blood transplant (UCBT).
Arm/Group | Umbilical Cord Blood Transplant
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplant (N=16)
Cardiac arrest (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 4 (5)
Encephalopathy (Nervous system disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Hepatobiliary disorders - Other, specify: VOD (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, specify: Adenovirus in plasma and adenovirus enteritis (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: BK virus infection with hemorrhagic cystitis (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: C.Difficile gastroenteritis (Infections and infestations) | 1 (1)
Infections and infestations - Other,specify:Hemorrhagic cystitis due to BK virus uremia and viremia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Sepsis without identified organism (Infections and infestations) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Nervous system disorders - Other, specify: Altered mental status (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify: Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory,thoracic and mediastinal disorders - Other,specify:Respiratory distress after sedation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory distress after sedation for PICC line rewiring
Sepsis (Infections and infestations) | 2 (2)
Vascular disorders - Other, specify: VOD (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplant (N=16)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Catheter related infection (Infections and infestations) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Infections and infestations - Other, specify: Adenovirus (Infections and infestations) | 1 (1)
Infections and infestations -Other,specify: Hemorrhagic cystitis due to BK virus uremia and viremia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Norovirus viral diarrheal disese (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Recurrent Clostridium Difficile colitis (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify: Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT01247701/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT01247701/ICF_000.pdf